CLINICAL TRIAL: NCT00951639
Title: Cassia Cinnamon and Acute Endurance Exercise for the Enhancement of Glucose Uptake in Healthy Young Women
Brief Title: Cassia Cinnamon for Glucose Uptake in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: BaylorU_Cassia_Women
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Insulin Resistance; Impaired Glucose Tolerance; Prediabetes
Keywords: Cassia; Cinnamon; Blood Glucose; Endurance exercise; Acute exercise; Overweight; Obesity; Women
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Prediabetic State; Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5g Cassia cinnamon (Experimental): Experimental treatment group
  Interventions: Dietary Supplement: Cassia cinnamon
- 50 minutes endurnace exercise (Active Comparator): Endurance exercise treatment known to influence blood glucose
  Interventions: Procedure: 50 minutes exercise
- 5g Cellulose (Placebo Comparator): Placebo equivalent in weight and appearance to experimental treatment
  Interventions: Dietary Supplement: Cellulose Powder

INTERVENTIONS:
Dietary Supplement: Cassia cinnamon — 5g encapsulated ground bark administered once in experimental session
  Other Names: Brand: Nature's Bounty
  Arms: 5g Cassia cinnamon
Procedure: 50 minutes exercise — 50 minutes treadmill endurance exercise at 70% of the heart rate reserve (correlated to VO2max)
  Arms: 50 minutes endurnace exercise
Dietary Supplement: Cellulose Powder — 5g encapsulated powder administered during placebo experimental session
  Arms: 5g Cellulose

SUMMARY:
The purpose of this study was to compare the acute effects of 5g of Cassia cinnamon, 50 minutes of endurance exercise performed at 70% of the heart rate reserve (correlated to VO2max), and 5g of cellulose placebo on blood glucose, serum insulin and insulin sensitivity following an oral glucose tolerance test 3 hours after administration of each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* BMI: 27-45
* DXA body fat % greater than 30%
* 18-30 years of age
* Healthy
* From the Baylor University campus and surrounding community
* Regular sleep habits

Exclusion Criteria:

* Not regular users of any species of cinnamon
* Not diagnosed with any metabolic disorder or chronic medical condition
* Not taking prescription medications for 2 months before the study
* Not taking ergogenic aids for 2 months before the study
* Not taking oral contraceptives for 2 months before the study
* No IUD placed for 2 months before the study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | Baseline, 0, 30, 60, 90 and 120 minutes following OGTT

SECONDARY OUTCOMES:
Serum Insulin | Baseline, 0, 30, 60, 90 and 120 minutes following OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Darryn S Willoughby, Ph.D., Study Chair — Baylor University; Jean L Gutierrez, Ph.D., Principal Investigator — Baylor University
Locations (1):
- Baylor University Department of Health, Human Performance, and Recreation, Waco, Texas, United States

REFERENCES:
- [Background] Hlebowicz J, Darwiche G, Bjorgell O, Almer LO. Effect of cinnamon on postprandial blood glucose, gastric emptying, and satiety in healthy subjects. Am J Clin Nutr. 2007 Jun;85(6):1552-6. doi: 10.1093/ajcn/85.6.1552. PMID 17556692
- [Background] Hlebowicz J, Hlebowicz A, Lindstedt S, Bjorgell O, Hoglund P, Holst JJ, Darwiche G, Almer LO. Effects of 1 and 3 g cinnamon on gastric emptying, satiety, and postprandial blood glucose, insulin, glucose-dependent insulinotropic polypeptide, glucagon-like peptide 1, and ghrelin concentrations in healthy subjects. Am J Clin Nutr. 2009 Mar;89(3):815-21. doi: 10.3945/ajcn.2008.26807. Epub 2009 Jan 21. PMID 19158209
- [Background] Solomon TP, Blannin AK. Changes in glucose tolerance and insulin sensitivity following 2 weeks of daily cinnamon ingestion in healthy humans. Eur J Appl Physiol. 2009 Apr;105(6):969-76. doi: 10.1007/s00421-009-0986-9. Epub 2009 Jan 22. PMID 19159947
- [Background] Solomon TP, Blannin AK. Effects of short-term cinnamon ingestion on in vivo glucose tolerance. Diabetes Obes Metab. 2007 Nov;9(6):895-901. doi: 10.1111/j.1463-1326.2006.00694.x. PMID 17924872